CLINICAL TRIAL: NCT01339364
Title: Evaluation of Three 1-day Educational Intervention to Promote Knowledge and Attitude of Community Pharmacists About Evidence-based Weight Management
Brief Title: Impact of Three Continuing Education Meetings for Community Pharmacists on Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Kheirollah Gholami M.Sc., PharmD, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 240/4402
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Continuing Pharmacy Education; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Didactic Lecture (Active Comparator)
  Interventions: Other: Didactic Lecture
- Lecture plus Case Disscussion (Experimental)
  Interventions: Other: Interactive Lecture
- Lecture plus Small Group Education (Experimental)
  Interventions: Other: Lecture plus Small Group Education

INTERVENTIONS:
Other: Didactic Lecture — 2 sessions of didactic lecture with PowerPoint presentations each delivered by a special lecturer. whole education period lasts 3 hours.
  Arms: Didactic Lecture
Other: Interactive Lecture — 2 sessions of brief interactive lectures followed by case discussion sections.
  Arms: Lecture plus Case Disscussion
Other: Lecture plus Small Group Education — A 1.5 hours session of didactic lecture followed by a session of small group education with 3 simulated patients.
  Arms: Lecture plus Small Group Education

SUMMARY:
This study is a three-arm randomized controlled trial to evaluate the effects of 1-day continuing educational meetings for community pharmacists with three distinct educational methods: 1) Didactic lecture 2) Didactic lecture plus case discussion in a large group 3) Didactic lecture plus small group education with simulated patient

Knowledge and attitude of the participants would be measured as the study outcome in three periods: pre-education, post-education and 1 month after the meetings.

DETAILED DESCRIPTION:
The study is designed as an Instructor blinded-Randomized Controlled Trial.

An educational need assessment is undergone prior to educational content preparation by interviewing 5 community pharmacists. After educational content preparation by instructors, the outcome assessment tool (knowledge, attitude questionnaire) would be designed by a distinct investigator. Closed and Open-ended questions are included to investigate different levels of Bloom's taxonomy.

The questionnaire would be validated by specialists other than the instructors and it will piloted to investigate the reliability( Cronbach's Alfa > 0.7).

Community pharmacists of Tehran,Capital city of Iran, would be invited to participate in the study. The participants would be randomly assigned to 3 groups by random number table. Each group receives the same education content with a different method:

1. Didactic lecture
2. Didactic lecture plus case discussion in a large group
3. Didactic lecture plus small group education with simulated patient(SP). Interviewing with SP is conducted by small group facilitators with Brain Storming Technic.

Each participant receives a compact disk which includes the educational material and he/she would be able to contact the instructors by phone or e-mail during the follow-up period. (Reinforcement Phase)

ELIGIBILITY:
Inclusion Criteria:

* Community Pharmacist

Exclusion Criteria:

* Less than four hours of daily work in community pharmacy

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Knowledge Grade Points and Attitudes(Phase 1) | One day
  Obtained through a validated knowledge and attitude questionnaire.
Knowledge Grade Points and Attitudes(Phase 2) | One month(average of 4 weeks after the day of training)
  Obtained through a validated knowledge and attitude questionnaire.

SECONDARY OUTCOMES:
Satisfaction of Participants | One day
  Obtained by a Satisfaction Evaluation Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kheirollah Gholami, M.Sc, PharmD, Study Chair — Tehran University of Medical Sciences; Arash Rashidian, MD, PhD, Principal Investigator — Tehran University of Medical Sciences; Mohammadreza Javadi, PharmD, BCPS, Principal Investigator — Tehran University of Medical Sciences; Amir Sarayani, PharmD, MPH, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Faculty of Pharmacy-Tehran University of Medical Sciences, Tehran, Tehran Province, Iran